CLINICAL TRIAL: NCT07208578
Title: Non-invasive Hemodynamic Monitoring in COPD Patients Admitted to the Respiratory Intensive Care Unit: Reliability, Clinical Utility, and Ventilation-related Hemodynamic Changes
Brief Title: Prospective Evaluation of Electrical Cardiometry for Hemodynamic Monitoring in COPD Patients Admitted to the Respiratory Intensive Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousef Tharwat Geris Qrqar, resident at the Chest Diseases and Tuberculosis Department, Assiut University
Other Study IDs: Non-invasive Hemodynamic
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Non-invasive Electrical Cardiometry
Keywords: non-invasive electrical cardiometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Invasive Mechanical Ventilation Arm: COPD patients requiring intubation and invasive ventilation support. Hemodynamics will be continuously monitored using ICON to evaluate changes under invasive ventilation physiology.
- Non Invasive Mechanical Ventilation Arm: COPD patients managed with NIV (e.g., BiPAP/CPAP). The arm will assess ICON's ability to track hemodynamic responses to positive pressure without intubation.
- No Mechanical Ventilation Arm: COPD patients receiving supplemental oxygen therapy or room air only. This group serves as a baseline to study hemodynamic changes without ventilatory support.

SUMMARY:
This study investigates the reliability and clinical usefulness of non-invasive electrical cardiometry (ICON® device) in monitoring hemodynamic changes in COPD patients admitted to the respiratory intensive care unit (RICU).

DETAILED DESCRIPTION:
hemodynamic monitoring is critical in critically ill patients, especially those with COPD experiencing acute respiratory failure. Traditional invasive methods such as pulmonary artery catheterization are accurate but carry procedural risks. The ICON® device enables real-time, continuous, non-invasive assessment of parameters like cardiac output, stroke volume, systemic vascular resistance, and thoracic fluid content using thoracic bioimpedance. This prospective observational study will assess its reliability against clinical outcomes and evaluate the influence of different ventilation strategies (invasive, non-invasive, no ventilation) on hemodynamic changes. Data will be collected serially throughout ICU stay to determine ICON's contribution to optimizing patient management and risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Admission to RICU with COPD or COPD-related acute respiratory failure

Informed consent provided by patient or legal representative

Exclusion Criteria:

* patients <18 years

Pregnant women

Injuries, burns, or skin conditions preventing electrode placement

Patients with uncontrolled seizures

Patients needing electrical DC shock

Refusal or withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) admitted with a confirmed diagnosis of COPD or COPD-related acute respiratory failure requiring ICU admission. Patients may present with hypoxemia, hypercapnia, or both. Participants will include both male and female patients admitted for exacerbations or decompensation, receiving either invasive mechanical ventilation, non-invasive mechanical ventilation, or supplemental oxygen. Exclusions include patients with electrode placement limitations (e.g., skin injuries), seizure disorders, pregnancy, or those refusing consent.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac output (CO) measured by the electrical cardiometer (ICON®) in COPD patients admitted to the respiratory ICU. | Baseline
  The change in cardiac output values during the ICU stay as measured non-invasively by the ICON device, reflecting hemodynamic status.